CLINICAL TRIAL: NCT07223866
Title: The Impact of Physiologic Cataract Surgery on Patient Comfort and Medication Usage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew Rauen (Other)
Responsible Party: Sponsor-Investigator, Matthew Rauen, Principal Investigator, Wolfe Eye Clinic
Organization: Wolfe Eye Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IIT #98621123
Record Dates: First submitted 2025-10-20; First posted 2025-11-03 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Cataract and IOL Surgery; Cataract Surgery Anesthesia; Cataract Surgery Experience; Nuclear Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Study treatment & Methods:
  * Sequential cataract surgery with similar cataract grade 2-3+ based on LOCS III grading bilaterally; 2nd eye to be completed within 2-3 weeks of first eye
  * Randomize first eye to low vs high IOP, contralateral eye receives opposite IOP
  * Patient education on VAS with standard script
  * Standard pre-op drops: 2 drops of cyclopentolate 1%, tropicamide 1%, flurbiprofen sodium (Ocufen 0.03%), phenylephrine hydrochloride 2.5%, and 3 drops of marcaine 0.05%
  * After draping, patients receive OcuCoat on cornea and 3 drops of lidocaine, 1mg of Versed (midazolam for anxiety with no analgesic effects)
  * If patients experienced breakthrough pain during surgery, additional topical anesthetic, intracameral lidocaine, and/or opioid will be used per surgeon discretion and stage recorded
  * Physiological responses recorded: Anesthesiologist will monitor patients per standard of care but will record additional BP/HR values at the start of the case (room entry), 4 minutes
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Centurion with Active Sentry at a traditionally high IOP setting (Active Comparator): Centurion with Active Sentry at a traditionally high IOP setting, Eyes in this arm will maintain an Intraocular Pressure (IOP) of 65 millimeters of mercury (mmHg) throughout the cataract surgery.
  Interventions: Device: High IOP Setting
- Unity VCS/CS with Intelligent Fluidics at a low IOP setting (Active Comparator): Unity VCS/CS with Intelligent Fluidics at a low IOP setting. Eyes in this arm will maintain an Intraocular Pressure (IOP) of 25 millimeters of mercury (mmHg) throughout the cataract surgery.
  Interventions: Device: Low IOP Setting

INTERVENTIONS:
Device: High IOP Setting — Prospective, single-surgeon, eyes undergoing phacoemulsification will be randomized to low (IOP 25mmHg) or high (IOP 65mmHg) IOP, contralateral eye will receive other treatment
  Arms: Centurion with Active Sentry at a traditionally high IOP setting
Device: Low IOP Setting — Prospective, single-surgeon, eyes undergoing phacoemulsification will be randomized to low (IOP 25mmHg) or high (IOP 65mmHg) IOP, contralateral eye will receive other treatment
  Arms: Unity VCS/CS with Intelligent Fluidics at a low IOP setting

SUMMARY:
The study will pertain to investigating the impact of high vs low IOP on the intraoperative experience and comfort for the patient and surgeon. Our hypothesis is that operating at a more physiological IOP using Unity VCS/CS and Centurion with Active Sentry at a higher, or more traditional IOP will result in significantly less discomfort/pain as assessed by the decreased need for rescue medication and lower VAS scores.

DETAILED DESCRIPTION:
Objective/ Unmet Medical Need:

To investigate the impact of Unity VCS/CS with Intelligent Fluidics at a low IOP setting and Centurion with Active Sentry at a traditionally high IOP setting on the intraoperative experience for the patient and surgeon. Limited research on phacoemulsification at near physiological IOP and its impact on patient discomfort/pain using the Unity VCS/CS system.

Design:

Prospective, single-surgeon, eyes undergoing phacoemulsification will be randomized to high (IOP 65mmHg) or low (IOP 25mmHg) IOP, contralateral eye will receive other treatment.

STUDY HYPOTHESIS Unity VCS/CS with Intelligent Fluidics during cataract surgery will result in significantly less discomfort/pain as assessed by the decreased need for rescue medication and lower VAS scores.

ELIGIBILITY:
Inclusion Criteria: Subjects who will require bilateral cataract surgery will be considered. Evaluations will occur in the clinic of the Principal Investigator (PI) Matthew Rauen, MD at the Wolfe Eye Clinic.

Inclusion Criteria:

* Visually significant cataract 2-3+ undergoing uncomplicated cataract surgery with similar cataract grade in both eyes
* Unremarkable ocular health but inclusive of early AMD

Exclusion Criteria:

* H/o ocular surgery including corneal refractive surgery
* Compromised zonular integrity or stability
* Uncontrolled diabetes and diabetic retinopathy
* Small pupils
* H/o systemic inflammatory disease/uveitis
* H/o chronic pain medications (including narcotics) and benzodiazepine usage
* Abnormal liver or renal function

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Rescue Medication | During cataract surgery
  Percent of pts in each group requiring rescue medication for breakthrough discomfort/pain

SECONDARY OUTCOMES:
VAS Pain Score | During Phaco, I/A, and Visco Removal
  Discomfort/pain score at phaco, I/A, visco removal. VAS score : 0 - no pain, 10 - unbearable pain
Surgeon Intraoperative Experience | During cataract surgery
  1- Poor: fluctuating chamber (reverse pupillary block or surge) and reduced efficiency (nucleus & cortex removal)
  * 2- Good: >75% chamber stability and adequate efficiency
  * 3- Excellent: Minimal to no fluctuating chamber and excellent efficiency
Cost Analysis | During cataract surgery
  Cost-analysis on intraoperative medications utilized in high vs low IOP groups
Breakthrough pain and discomfort High Axial Length | During cataract surgery
  VAS Pain score on subjects with axial length of >24.5mm VAS score : 0 - no pain, 10 - unbearable pain If patients experienced breakthrough pain during surgery, additional topical anesthetic, intracameral lidocaine, and/or opioid will be used per surgeon discretion and stage of surgery recorded.
1 day Post Op Patient Survey | 1 day post op cataract surgery, each eye
  * on experience (Iowa Satisfaction with Anesthesia Scale (ISAS)
  * on patient preference - What eye was more comfortable? (R/L)
  * surgical experience did you enjoy more? (R/L)
  * x% of eyes would undergo the same procedure again
  * x% of eyes would recommend the procedure to family and friends
Anesthesiologist Review Blood Pressure | During cataract surgery
  Physiological responses recorded: Anesthesiologist will monitor patients per standard of care but will record additional Blood Pressure values at the start of the case (room entry), 4 minutes after versed is administered, during phacoemulsification, and during viscoelastic removal.
Anesthesiologist Review Pulse Rate | During cataract surgery
  Physiological responses recorded: Anesthesiologist will monitor patients per standard of care but will record additional Pulse Rate values at the start of the case (room entry), 4 minutes after versed is administered, during phacoemulsification, and during viscoelastic removal.

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfe Eye Clinic and Wolfe Surgery Center, West Des Moines, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share informed consent and study protocol.
Supporting Information: Study Protocol, ICF
Time Frame: Will provide with this submission.
Access Criteria: No patient specific data analysis will be shared. Will supply copies of IRB approved informed consent and protocol. Inquires to be sent to rkohler@wolfeclinic.com

REFERENCES:
- [Background] Liu YC, Setiawan M, Ang M, Yam GHF, Mehta JS. Changes in aqueous oxidative stress, prostaglandins, and cytokines: Comparisons of low-energy femtosecond laser-assisted cataract surgery versus conventional phacoemulsification. J Cataract Refract Surg. 2019 Feb;45(2):196-203. doi: 10.1016/j.jcrs.2018.09.022. Epub 2018 Dec 6. PMID 30528516
- [Background] Scarfone HA, Rodriquez EC. Evaluation of Early Changes of the Anterior Vitreous Interface after Cataract Surgery, using Low-Pressure Settings Determined by OCT. ASCRS 2023 May 6, San Diego Convention Center. https://ascrs.confex.com/ascrs/23am/meetingapp.cgi/Paper/88373
- [Background] Donnenfeld ED, Mychajlyszyn D, Mychajlyszyn A, Stein R. Pain control and reduction of opioid use associated with intracameral phenylephrine1.0%-ketorolac 0.3% administered during cataract surgery. J Cataract Refract Surg. 2022 Jul 1;48(7):759-764. doi: 10.1097/j.jcrs.0000000000000855. Epub 2021 Oct 29. PMID 34860481
- [Background] Reddy AJ, Dang A, Dao AA, Arakji G, Cherian J, Brahmbhatt H. A Substantive Narrative Review on the Usage of Lidocaine in Cataract Surgery. Cureus. 2021 Oct 30;13(10):e19138. doi: 10.7759/cureus.19138. eCollection 2021 Oct. PMID 34737914
- [Background] Crandall AS, Zabriskie NA, Patel BC, Burns TA, Mamalis N, Malmquist-Carter LA, Yee R. A comparison of patient comfort during cataract surgery with topical anesthesia versus topical anesthesia and intracameral lidocaine. Ophthalmology. 1999 Jan;106(1):60-6. doi: 10.1016/S0161-6420(99)90007-6. PMID 9917782
- [Background] Gills JP, Cherchio M, Raanan MG. Unpreserved lidocaine to control discomfort during cataract surgery using topical anesthesia. J Cataract Refract Surg. 1997 May;23(4):545-50. doi: 10.1016/s0886-3350(97)80211-8. PMID 9209989

DOCUMENTS (2):
  • Study Protocol (2025-10-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT07223866/Prot_000.pdf
  • Informed Consent Form (2025-10-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT07223866/ICF_001.pdf